CLINICAL TRIAL: NCT06780423
Title: Structural Characteristics of Trunk and Limb Muscles in Cachectic Colorectal Cancer Patients
Acronym: CTLm-CCP
Status: Recruiting | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, prof. dr. Kenneth Verboven, Prof. dr., Hasselt University
Other Study IDs: 2021/148 - CTLm-CCP
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer; Cancer Cachexia
Keywords: colorectal cancer; cachexia; skeletal muscle; skeletal muscle fibers; capillarization
MeSH Terms: conditions — Colorectal Neoplasms; Cachexia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples With DNA — * muscle biopsies
  * blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cachectic colorectal cancer patients
  Interventions: Procedure: Minimal invasive fine needle muscle biopsies
- Non-cachectic colorectal cancer patients
  Interventions: Procedure: Minimal invasive fine needle muscle biopsies
- Healthy controls
  Interventions: Procedure: Minimal invasive fine needle muscle biopsies

INTERVENTIONS:
Procedure: Minimal invasive fine needle muscle biopsies — Fine needle muscle biopsies will be taken from the m. erector spinae and the m. vastus lateralis. Participants are placed in a standardized prone position on the examination table for measurements of the m. erector spinae and in a supine position for measurements of the m. vastus lateralis.

SUMMARY:
Until now, cancer is still associated with high morbidity and mortality, and is therefore a big issue for the public health. Colorectal cancer is the second leading cause of cancer death in developed countries. In advanced colorectal cancer, 60% of these patients develop cachexia. The presence of cachexia plays an important role in the high mortality rate of cancer. Cachexia is characterized by involuntary weight loss with loss of skeletal muscle with or without loss of fat mass.

The aim of this study is to determine the feasibility of taking muscle biopsies of cachectic colorectal cancer patients. Skeletal muscle characteristics will be compared between biopsies of the m. erector spinae and the m. vastus lateralis from cachectic colorectal cancer patients, non-cachectic colorectal cancer patients and healthy controls.

10 cachectic, 25 non-cachectic, and 25 healthy controls will be recruited for this study. It is an observational study, so measurements will be taken at one time point. Interventions/measurements:

* muscle biopsies
* blood samples
* 3D freehand ultrasound
* Short physical performance battery test
* handgrip strength
* questionnaires (activity pattern, quality of life)

ELIGIBILITY:
Cachectic colorectal cancer patients.

Inclusion criteria:

* minimum age of 18 years old
* unwanted weight loss > 5% in the last 6 months OR > 2% unwanted weight loss in combination with a BMI < 20kg/m2 OR >2% unwanted weight loss in combination with sarcopenia
* Cachexia staging score (CSS): 5-12

Exclusion Criteria:

* Mental of psychological condition
* Insufficient knowledge of the Dutch language
* Muscle diseases affecting the spine and lower limbs
* Bedridden

Non-Cachectic cancer patients.

Inclusion criteria:

* minimum age of 18 years old
* No unwanted weight loss > 5% in the last 6 months OR > 2% unwanted weight loss in combination with a BMI < 20kg/m2 OR >2% unwanted weight loss in combination with sarcopenia
* Cachexia staging score (CSS): 0-2

Exclusion criteria:

* Mental of psychological condition
* Insufficient knowledge of the Dutch language
* Muscle diseases affecting the spine and lower limbs
* Bedridden

Healthy controls.

Inclusion criteria:

- minimum age of 18 years old

Exclusion criteria:

* Mental of psychological condition
* Insufficient knowledge of the Dutch language
* Muscle diseases affecting the spine and lower limbs
* Bedridden

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 12 cachectic colorectal cancer patients, 25 non-cachectic colorectal cancer patients, and 25 healthy controls will be recruited in the study. Colorectal cancer patients will be recruited by the surgeans from the Jessa Hospital (Hasselt, Belgium), and the healthy controls will be recruited by the local researcher from Hasselt University.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-23 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle fiber typing | at enrollment
  Immunofluorescence staining of skeletal muscle biopsies to observe different muscle fiber types (myosin heavy chains)
skeletal muscle nuclei | at enrollment
  Immunofluorescence staining with DAPI
Inflammatory parameters | at enrollment
  ELISA (bloodsamples), immunofluorescence staining (muscle biopsies)
Mitochondrial morphology | at enrollment
  mitochondrial fusion and fission (western blot) mitochondrial OXPHOS (western blot)

SECONDARY OUTCOMES:
3D freehand ultrasound | at enrollment
  measuring the volume of the m. rectus femoris
CT-scans | at enrollment
  level lumbar 3 To calculate the cross-sectional area of the m. erector spinae.
Activity pattern | at enrollment
  PASIPD questionnaire
VAS score | at enrollment
  to descripe the pain at the moment of the biopsy procedure. Score range is 0 to 10. With 0 no pain until 10 the worst pain.
Handgrip strength | at enrollment
  Using the JAMAR to measure the handgripstrength
Short Physical Performance Battery (SPPB) test | at enrollment
  Including a balance test, sit-to-stand test and four meter walking test
Quality of Life questionnaire | at enrollment
  SF-36 questionnaire
  36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
skeletal muscle capillarization | at enrollment
  Immunofluorescence staining for capillaries in the skeletel muscle biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Verboven, Professor, Principal Investigator — Hasselt University - REVAL
Locations (2):
- Belgium (2):
  - Hasselt University - REVAL research institution, Diepenbeek, Limburg
  - Jessa Hospital, Hasselt, Limburg